CLINICAL TRIAL: NCT06626230
Title: An Incremental Dose Escalation Trial of Safety and Tolerability of Curcumin
Brief Title: Safety of Anal Curcumin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lisa Flowers (Other)
Responsible Party: Sponsor-Investigator, Lisa Flowers, Professor, Emory University
Organization: Emory University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007193
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Anal High Grade Squamous Intraepithelial Lesion
Keywords: HSIL/AIN 2-3; Curcumin; Cancer; Human Papillomavirus (HPV); HIV; Curcuminoids
MeSH Terms: conditions — Neoplasms | interventions — Diarylheptanoids; turmeric extract; Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Level 1 (Experimental): Participants will receive a supply of curcumin gelatin capsules to insert 500 mg intra-anally every day for a 14-day treatment period
  Interventions: Drug: Curcuminoid Capsules
- Dose Level 2 (Experimental): Participants will receive a supply of curcumin gelatin capsules to insert 1000 mg intra-anally every day for a 14-day treatment period
  Interventions: Drug: Curcuminoid Capsules
- Dose Level 3 (Experimental): Participants will receive a supply of curcumin gelatin capsules to insert 1500 mg intra-anally every day for a 14-day treatment period
  Interventions: Drug: Curcuminoid Capsules
- Dose Level 4 (Experimental): Participants will receive a supply of curcumin gelatin capsules to insert 2000 mg intra-anally every day for a 14-day treatment period
  Interventions: Drug: Curcuminoid Capsules
- Dose Level 5 (Experimental): Participants will receive a supply of curcumin gelatin capsules to insert 2500 mg intra-anally every day for a 14-day treatment period
  Interventions: Drug: Curcuminoid Capsules
- Dose Level 6 (Experimental): Participants will receive a supply of curcumin gelatin capsules to insert 3000 mg intra-anally every day for a 14-day treatment period
  Interventions: Drug: Curcuminoid Capsules
- Dose Level 7 (Experimental): Participants will receive a supply of curcumin gelatin capsules to insert 3500 mg intra-anally every day for a 14-day treatment period
  Interventions: Drug: Curcuminoid Capsules
- Dose Level 8 (Experimental): Participants will receive a supply of curcumin gelatin capsules to insert 4000 mg intra-anally every day for a 14-day treatment period
  Interventions: Drug: Curcuminoid Capsules

INTERVENTIONS:
Drug: Curcuminoid Capsules — 500 mg curcuminoids from C3 Complex capsule. Curcuma longa (Turmeric), a constituent of the spice turmeric, is considered a low-toxicity, dietary-derived agent with chemopreventive and therapeutic benefits Study participants will be instructed to insert the curcumin capsules gelatin intra-anally every day for a 14-day treatment period.
  Escalating doses
  Other Names: Curcumin C3 Complex; Curcuma longa (Turmeric)

SUMMARY:
The purpose of this study is to see if curcumin can reverse anal high-grade squamous intraepithelial lesions (aHSIL) (high-grade anal precancerous cells or high-grade abnormal cells) in people living with HIV to avoid current treatments such as ablation (destroying abnormal cells with heat or surgical excision (cutting out the abnormal cells)), which have potential short- and long-term side effects.

DETAILED DESCRIPTION:
This proposal suggests conducting a Phase I clinical trial using a 3 + 3 dose escalation approach to assess the safety and determine the maximum tolerated dose of intra-anal curcumin in individuals with HIV who have anal high-grade squamous intraepithelial lesions (aHSIL/AIN 2-3). Currently, there is a significant need for non-surgical treatments for pre-malignant anal diseases in people with HIV, aiming to reduce risks and complications associated with existing surgical and topical interventions.

Curcumin, a compound derived from turmeric, is known for its anti-inflammatory and anti-infectious properties. While previous research has shown its anticancer effects in oral doses, its bioavailability is limited, and intra-anal administration has not been studied in humans. This trial aims to explore the potential of intra-anal curcumin as an alternative treatment for aHSIL in people with HIV.

The study will involve enrolling participants with aHSIL and administering increasing doses of curcumin intra-anally for 14 days, following the 3 + 3 dose escalation model. The trial will continue until the dose-limiting toxicity (DLT) level is reached, and participants report symptoms necessitating a dose reduction.

To enhance future studies, the researchers will also evaluate patient and male partner acceptability through questionnaires. The insights gained from this trial will guide the design of subsequent efficacy and safety studies for individuals with AIN 2 and 3 neoplasia.

ELIGIBILITY:
Major Inclusion Criteria:

* 30 and older
* Have biopsy-proven anal intraepithelial neoplasia (AIN) 2, AIN 3 without previous treatment
* Or cytology results for ASC-H or HSIL
* Able and willing to complete Study Diary
* Other inclusion criteria apply

Exclusion Criteria:

* Have a clinically significant chronic medical condition that is considered progressive, such as but not limited to coronary disease, congestive heart failure, chronic obstructive lung disease, and diabetes mellitus. Chronic nonprogressive or intermittent syndromes are not excluded, including migraine headaches, mild reactive airway disease, controlled hypertension, stable pain syndromes, or benign gastric reflux.
* Have any history of anal cancer malignancy.
* Pregnant or planning to become pregnant in the next three months.
* Have a history of sensitivity or allergy to any compound used in this study.
* Have Grade 2 or higher renal or hematology abnormality,
* Are currently using, or in the last year have used intravenous drugs (except for therapeutic use), recreational drugs, or alcohol abuse.
* Other exclusion criteria apply

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Maximum curcumin tolerated dose | Up to 22 days after treatment
  To determine the maximum tolerated dose (MTD) of curcumin, toxicities will be tabulated and reported per dose level according to grade and type of toxicity experienced. The dose level at which no more than 33% of study participants have a DLT will be considered the maximum tolerated dose.

SECONDARY OUTCOMES:
Toxicity related to treatment | Up to 22 days after treatment
  Toxicities will be tabulated and reported per dose level according to grade and type of toxicity experienced (tolerability of curcumin). Participants will be monitored during the trial for adverse events, tolerability, and compliance using the Common Terminology Criteria for Adverse Events (CTCAE). Side effects will be recorded in a study diary maintained by the participant.
Anoscopy changes | 22 days after treatment
  Participants will receive an anoscopy to examine the anus and perineum for any findings outlined in the anoscopic findings chart (Safety of curcumin intra-anal powder)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, MD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Grady Hospital - Ponce De Leon Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified Individual participant data that underlie the published results will be made available for sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available from December 2025 to January 2031.
Access Criteria: Data will be available for sharing with researchers providing a methodologically sound proposal, to achieve aims in the approved proposal. Proposals should be directed to lflowe2@emory.edu. The data requestor needs to sign a data access agreement to gain access.